CLINICAL TRIAL: NCT06000631
Title: Short-term and Long-term Effectiveness of Different Dosage Parameters in Looking Behaviors, Functional Skills and Caregiver-child Interaction of Early Powered Mobility Training for Toddlers With Motor Delays
Brief Title: Long-term Effectiveness of Different Dosage Parameters of Early Powered Mobility Training for Toddlers With Motor Delays
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Han Huang, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112WFD2610076
Record Dates: First submitted 2023-07-03; First posted 2023-08-21 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Young Children With Motor Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-hour session of ROC-Stand training for a total of 48 hours (ROC-Stand(2-hr)) (Active Comparator): A licensed, independent therapist and caregivers will provide the training program in the public space in the university for 2 hours/per session, 2 sessions/per week for a total of 12-week intervention based on ecological and dynamic systems theories. Each week the participant will wear a light-weight, head-mounted eye-tracker for recording the first 10-minute of driving and natural play sessions in a 2-hour training session. The 2-hour training session is composed of a 70-minute driving session and a 50-minute natural play session. Training will concentrate on building the concept of casual-effect on the control system and car motion, practicing goal-oriented driving in certain public spaces, upper limb use in functional tasks for exploration in driving sessions, and applying various motor skills for mobility and socialization in natural play sessions. The program will be discussed by the family and the treating therapist.
  Interventions: Behavioral: Ride-On Car Training in a standing posture with a 2-hour session
- 1-hour session of ROC-Stand training for a total of 48 hours (ROC-Stand(1-hr)) (Active Comparator): The same therapist for the ROC-Stand(2-hr) group will be responsible for the program. The training frequency and guidelines are the same as the ROC-Stand(2-hr) group, except for the training intensity of 1-hour per session and intervention duration for 24 weeks. Each 1-hour session will include a 35-minute car play and a 25-minute natural play. The participants will also wear the head-mounted eye tracker in one training session for recording 20 minutes (the first 10-minute of driving and the first 10-minute of natural play) every week.
  Interventions: Behavioral: Ride-On Car Training in a standing posture with a 1-hour session
- 1-hour session of conventional therapy for a total of 48 hours (Control(1-hr)) (Active Comparator): Another licensed, independent therapist will provide the training program to the Control(1-hr) group for 1 hours/per session, 2 sessions/per week for a total of 24-week intervention. The conventional therapy provided in the Control(1-hr) group is based on the developmental and motor learning theories. The goals are to improve certain motor skills or psychosocial skills based on each participant's current developmental stage. The general propose of the training is to facilitate the developmental scales and improve certain mobility, socialization and upper limb use in functional tasks. Each participant will have the opportunity to walk on the same public space as the ROC training groups and interact with the therapist and caregivers depending on his/her motor abilities. The participants will also wear the head-mounted eye-tracker for the first 20 minutes in one training session every week.
  Interventions: Behavioral: Conventional Therapy with a 1-hour session

INTERVENTIONS:
Behavioral: Ride-On Car Training in a standing posture with a 2-hour session — A licensed, independent therapist and caregivers will provide the training program in the public space in the university for a total of 12-week intervention based on ecological and dynamic systems theories. Training will concentrate on building the concept of casual effect on the control system and car motion, practicing goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person, play hide-and-seek) in certain public spaces, including hallways, convenient stores, garden, museum and upper limb use in functional tasks with driving, facilitating hand use in functional tasks for exploration and applying various motor skills for mobility and socialization in natural play session. Every week's treatment program will preplanned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Participants will continue their regular therapy during the whole study.
  Other Names: ROC-Stand(2-hr)
  Arms: 2-hour session of ROC-Stand training for a total of 48 hours (ROC-Stand(2-hr))
Behavioral: Ride-On Car Training in a standing posture with a 1-hour session — A licensed, independent therapist and caregivers will provide the training program in the public space in the university for a total of 24-week intervention based on ecological and dynamic systems theories. Training will concentrate on building the concept of casual effect on the control system and car motion, practicing goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person, play hide-and-seek) in certain public spaces, including hallways, convenient stores, garden, museum and upper limb use in functional tasks with driving, facilitating hand use in functional tasks for exploration and applying various motor skills for mobility and socialization in natural play session. Every week's treatment program will preplanned and adjusted by the therapist and the caregivers through discussion and clinical observation of the participant's performance in the previous session. Participants will continue their regular therapy during the whole study.
  Other Names: ROC-Stand(1-hr)
  Arms: 1-hour session of ROC-Stand training for a total of 48 hours (ROC-Stand(1-hr))
Behavioral: Conventional Therapy with a 1-hour session — The other independent OT will be responsible for providing conventional therapy in the same location as the ROC-Stand training for a total of 24-week intervention based on the developmental and motor learning theories. The goals are to improve certain motor skills or psychosocial skills based on each participant's current developmental stage. The general purpose of the training is to facilitate the developmental scales and improve mobility, socialization, and upper limb use in functional tasks.
  Other Names: Control(1-hr)
  Arms: 1-hour session of conventional therapy for a total of 48 hours (Control(1-hr))

SUMMARY:
The three purposes of this study are: 1) to compare the effects on looking behaviors, visual fixation and social interaction through the use of a head- mounted, eye-tracker in toddlers with motor disabilities after receiving different intensity levels of ROC-Stand training; 2) to compare short-term and long-term outcomes in terms of body function, activity and participation across the ICF framework, family perceptions and participation; and 3) to identify factors that predict individual differences in outcomes for toddlers with motor delays with the two dosing protocols. Based on the power analysis from the pilot study, the investigators will recruit 30 toddlers with motor delays and further randomly assign the participants to the 3 groups with the same total amount of 48-hour training, including 2 ROC-Stand groups and 1 conventional therapy group, i.e., an intensity level of 2-hour session of ROC-Stand training (ROC-Stand(2-hr)) (n=10), an intensity level of 1-hour session of ROC-Stand training (ROC-Stand(1-hr)) (n=10), and an intensity level of 1-hour session of conventional therapy (Control(1-hr)) (n=10). The training frequency for the 3 groups is 2 sessions/per week. The whole study duration will be 1 year. The head-mounted cameras worn by the participants will record the visual and interactive behaviors for 20 minutes/per week during intervention. Standardized assessments are provided for a total 4 times, including the time before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4). Assessments include body function, activity and participation across the ICF domains, family perception and participation. The findings of this study will provide guidelines for adjusting the dosage parameters of early powered mobility depending on each child's and family's needs.

DETAILED DESCRIPTION:
To evaluate the varying dosages' impact, the pilot RCT studied two different intensity levels of the ROC-Stand training for toddlers with motor delays. Initial findings suggest that the 48-hour regimen (2 hours per session, 2 sessions weekly) and the 24-hour approach (1 hour per session, 2 sessions weekly) have beneficial effects on the mobility and social functionalities of the toddlers. While enhancements were observed across the board during the 12-week intervention and follow-up phases, it was the ROC-48 group that showcased the most significant number of participants achieving clinically meaningful changes. This data implies that a 48-hour dose of ROC-Stand training may be the optimal requirement for noted improvements. Furthermore, another pilot study involving two participants using a lightweight, head-mounted eye-tracker by Positive Science, LLC during the ROC training phase has highlighted a positive trend in visual behaviors. Post-training, there was a noticeable increase in participants' interactions with their surroundings, particularly during social encounters and navigation. On the flip side, the frequency with which they observed faces and bodies reduced. The integration of eye-tracking technology showcases its potential in gauging participants' behaviors during self-initiated movements and interactions with the environment and caregivers. It offers a promising avenue to discern the type of visual and social cues acquired during early powered mobility training, aiding in comprehending environmental factors' influence on the psychosocial functions in toddlers with motor delays.

This study seeks to address the quest for determining the minimal effective dosage and to bolster its clinical utility in Taiwan. The research intends to contrast the effectiveness of two intensity levels of the ROC-Stand training, namely 2-hour and 1-hour sessions, targeting children aged between 1-3 at the outset of the intervention. With a 1-year follow-up, the study will not only provide insights into the ROC-Stand training but will also introduce a control group receiving the conventional 1-hour weekly therapy. To ensure consistency, each group will be subjected to the same frequency and duration, totaling 48 hours of intervention. This design of three-group comparison will enable us to define precise dosing benchmarks, incorporating a 2-hour ROC-Stand session (ROC-Stand(2-hr)), a 1-hour ROC-Stand session (ROC-Stand(1-hr)), and a 1-hour conventional therapy session (Control(1-hr)). Pinpointing these intensity benchmarks is vital for guiding clinical decisions and influencing health policy. In addition, the study's incorporation of a novel head-mounted eye-tracker, specifically tailored for young movers, anticipates capturing the nuances and diversities of real-world mobility interactions.

Method: This study will use a randomized, multi-group pretest-posttest control group design. Each group will undergo an intervention with a consistent frequency and duration, specifically, 2 sessions per week culminating in a total of 48 hours of training. The study will utilize a 3-group comparison structure, focusing on two distinct intensity levels. Building on previous research and the aims of this study, the three groups will be distinguished by the intensity of their respective training sessions: The ROC-Stand(2-hr) group will participate in 2-hour sessions twice a week for a total of 12 weeks (3 months). In contrast, both the ROC-Stand(1-hr) and Control(1-hr) groups will attend 1-hour sessions twice weekly for a period of 24 weeks (6 months).

Participants: The study will involve 30 toddlers aged between 12 to 36 months, all exhibiting motor delays. These participants will be randomly allocated to one of three groups: ROC-Stand(2-hr) (10 toddlers), ROC-Stand(1-hr) (10 toddlers), or Control(1-hr) (10 toddlers). Given the emphasis on early powered mobility training, the sample size determination hinges on an effect size f of 0.3, derived from preliminary PEDI-C mobility function data. With a power set at 0.8, a two-sided type I error rate of 0.05, anticipated 20~25% attrition, and drawing from recruitment patterns in past studies, the resulting requisite total sample size is estimated at 30 toddlers.

Recruitment: The participants will be recruited from self-referrals, health care practitioners, or the hospitals in Taoyuan or New Taipei where toddlers with motor delays are receiving outpatient rehabilitation. Children of parents/guardians who provide informed consent will participate in the study.

Procedure: Participants will undergo pre-intervention evaluations encompassing standardized developmental assessments, home environment and parental perception questionnaires. These will be administered by a licensed, independent OT, who is not participating in the training. Assessments will be conducted at four intervals: prior to training (T1), 3 months post-initiation (T2), 6 months post-initiation (T3), and a year after starting (T4). All participants will commence their training at the university. During the intervention, a lightweight head-mounted eye-tracker will record participants' eye gaze, manual actions, and social interactions once a week. An activity log, previously used in other studies, will document training conditions and caregiver feedback weekly. In the follow-up stage, participants will only attend their usual therapy sessions outside the study. Details of these sessions, including type, frequency, and dosage, will be documented at all four testing intervals. Undergraduate students will code the eye-tracking data. To ensure reliability, inter-rater scores will be calculated between these coders before the formal coding process begins.

Intervention:Two licensed occupational therapists who involve providing the training programs will ask caregivers to identify goals and measure progress using goal attainment scaling (GAS) at T1, T2, T3 and T4 time points for the 3 groups. The ROC-related programs require one therapist working with the caregivers based on the coaching technique described in the family-centered service model. The ROC involves a standing posture. The training principles are similar to those applied in the previous studies of ROC training in various environments. The conventional therapy program is a child-centered, therapist-directed program which is implemented by another therapist. Participants will have a necessary break depending on their endurance during training. In addition, all participants in the 3 groups will wear an eye-tracking headgear (Positive Science, LLC) to record the looking, fixation and interactive behaviors for one session/per week during intervention. All participants in the 3 groups will continue their regular therapy from their own clinics throughout the 1-year duration of the study, including physical therapy, occupational therapy, speech therapy, and other therapy.

Follow-up: This period will involve a follow-up phase following the above treatment programs; during this time no training programs will be delivered to the participants except for their own regular therapy.

Instrument and Procedure: To obtain the data of locomotor experience, an objective measure of using a head-mounted, eye-tracker and qualitative measures of activity logs will be applied during the intervention (training) phase. Standardized assessments as the quantitative measures will be administered at T1, T2, T3 and T4 in a testing room of the university. An independent, licensed OT who is blinded to the group assignment and study hypotheses will complete the assessments.

Descriptive statistics (frequency, means, standard deviations) of each behavior will be calculated. Kolmogorov-Smirnov will be used to examine whether the data follows a normal distribution. To compare the baseline characteristics of the major 3 groups, one way ANOVA (for data with normal distribution) and Kruskal-Wallis analysis of variance (for data with non-normal distribution) will be conducted. Data will be analyzed based on an intention-to-treat analysis. For those data collected during the intervention phase, descriptive statistics (frequency, means, standard deviations) of looking behaviors, visual fixation and interactive behaviors will be calculated and repeated measures analysis of variance will be used to compare the effects on each exploratory behaviors among the 3 training groups during intervention. A repeated measures analysis of variance (group [3] × time [4]) will be employed to evaluate the treatment effects on the secondary outcomes within and among the 3 groups at T1, T2, T3 and T4, followed by a post-hoc analysis using Bonferroni test to determine between which groups the differences occur. To clarify the relationship between other relevant factors and psychosocial outcomes, the investigators will consider two co-variates in the analysis based on previous research: motor composite scores from the Bayley-III and caregiver-child dysfunctional interaction (obtained from parenting stress index). Last, the investigators will apply a coefficient test for analyzing the relationship among the social function, looking/manual actions and social interactions, and caregiver-child dysfunctional interaction during the intervention phase in each group. SPSS 21.0 (SPSS Inc. Chicago, Illinois, USA) will be used for statistical analysis. Significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. age between 1-3 years old
2. motor delays that resulted in motor delays that prevented independent walking (> 1.5 standard deviation [SD] below the mean, assessed by the Chinese Child Development Inventory via a pediatric physician)
3. being able to stand independently for two seconds or tolerate standing with support for 10 minutes
4. being able to reach objects with either one or both hands
5. 69 to 103 cm height and 7 to 18 kg weight
6. parents agreeing to provide consent for their child's participation in the training program

Exclusion Criteria:

1. children with severe sensory impairments (including blindness or deafness)
2. exceeding the height or weight criteria
3. parents/guardians who are unable to make the time commitment for the program
4. children with severe emotional reactions which may result in harm

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Frequency of Looking and Fixation Behaviors at 24 weeks | 20 minutes/per week from the first week until the final week of intervention, up to 24 weeks
  Every week during the intervention phase, the first 10-minute of driving session and the first 10-minute of natural play session will be recorded from the eye-tracker for coding. The following behaviors will be coded, including looking behaviors (face, body, toy, environment and object looking) and fixation behaviors during different encounters (social, obstacle, manual and destinations).

SECONDARY OUTCOMES:
The Bayley Scales of Infant and Toddler Development-Third Edition (Bayley-III) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  an internationally recognized set of developmental tests with high reliability and validity applied to examine participants' developmental abilities. The Bayley has subsets of tests for motor, cognitive, and language development for children aged from 1 month to 42 months. It is a standardized assessment that can classify children's severity level of motor delays into four levels based on their motor composite scores, classified as severe (scores <55), moderate (55-69), mild (70-84), and no (>85) motor delays.
Infant/Toddler Sensory Profile - Chinese version (ITSP-C) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A standardized, norm-reference questionnaire of sensory processing ability in children at 0-3 years of age from caregiver's observations. Based on the criteria of age, the version for older children (7-36 months old) consisting of 48 item questions will be used in this study. The ITSP-C includes five sensory processing sections (Auditory, Visual, Vestibular, Tactile, and Oral Sensory Processing) and uses a 5-point Likert scale from 1 (almost always) to 5 (almost never). The ITSP-C with the Taiwanese norm has been established with good reliability and validity.
Peabody Developmental Motor Scales - Second edition (PDMS-2) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A norm referenced, standardized assessment of gross and fine motor skills in children 0-6 years. The PDMS-2 has been validated as a discriminative measure and demonstrated its' responsivity to change in infants and toddlers with cerebral palsy.
The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A caregiver's report questionnaire and five-point scale which measures both the instrumental and expressive aspects of mastery motivation. The DMQ involves seven subscales, including cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence. A higher score indicates higher motivation. For children aged 6 months to 19 years, the DMQ 18 previously showed good validity and reliability. Considering the age of participants, this study used two versions of the DMQ 18: infant's version (6-18 months) and preschooler's version (1.5-5 years).
The Chinese version of Pediatric Evaluation of Disability Inventory (PEDI-C) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A set of tests for children from 8 months to 6 years old. The PEDI-C quantifies self-care, mobility, and social function, and is particularly useful for tracking changes in functional skills. Each domain can be used separately for data analysis. The inter-rater and intra-rater reliabilities of the study reveal excellent agreement of the observations (0.95- 0.99), and good concurrent validity with the Functional Independence Measure for Children (Spearman ρ, 0.92-0.99).
Goal Attainment Scale (GAS) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A family-centered, criteria-referenced, responsive tool that includes five possible outcomes. A score of 0 indicates that the child has attained the goal, scores of -2 and -1 represent lower than expected performance, and +1 and +2 are higher than expected performance. It had good validity and excellent inter-rater agreements with ICCs of 0.90 or higher. The goals were incorporated into a single GAS composite score and converted to a T-score. A mean T-score of 50 indicated that the participants exceeded the expected level of goal performance.
The Chinese version of the Affordance in the Home Environment for Motor Development - Toddler version (AHEMDToddler-C) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese, Portuguese, and Spanish. Test-retest reliabilities for - Page 9 of 11 [DRAFT] - AHEMD-Toddler-C were adequate (0.46~0.93); for convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
The Parenting Stress Index Short Form (PSI/SF) | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A tool to measure measures the overall level of parenting stress experienced by parents/caregivers of children aged between one month and 12 years. The three subscales, that is, parental distress, parent-child dysfunctional interaction, and difficult child, add up to a total stress score. A higher score indicates higher stress. The PSI/SF is a tool with excellent validity and reliability.
Parental Perceptions | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  A set of questionnaires developed from the previous studies will be used at T1, T2 and T3 to examine parental perceptions on the PMDs use, the training programs and children's capabilities.
Activity Log | The test will be administered on four occasions: before training (T1), 3 months following initiation of training (T2), 6 months following initiation of training (T3), and the end of a year following initiation of training (T4)
  To record the training duration, locations, activities and the caregiver's feedback on the training program once every week during the intervention phase. The activity log will be mostly qualitative data that involves parents' descriptions

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Han Huang, ScD, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung University, Taoyuan, Taoyuan County
  - Linkou Chang Gung Memorial Hospital, Taoyuan, Taoyuan County